CLINICAL TRIAL: NCT02972788
Title: Effect of Enamel Matrix Proteins on Clinical Attachment Level and Alveolar Bone in Periodontal Maintenance Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0783-16-FB
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Periodontal Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — enamel matrix proteins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Group will receive enamel matrix protein derivative treatment along with scaling and root planing.
  Interventions: Drug: Enamel Matrix Proteins Derivative
- Control Group (Sham Comparator): Group will receive placebo (saline) treatment along with scaling and root planing.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Enamel Matrix Proteins Derivative — Enamel matrix proteins derivative will be placed in deep periodontal pocket during routine periodontal maintenance therapy.
  Other Names: Emdogain
  Arms: Experimental Group
Other: Saline — Saline will be placed in deep periodontal pocket during routine periodontal maintenance therapy.
  Arms: Control Group

SUMMARY:
The purpose of the study is to determine the effect of enamel matrix protein derivative on an inflamed, periodontal-involved tooth. The hypothesis to be studied is that enamel matrix derivative protein with increase the clinical attachment level is localized sites of advanced periodontal disease.

DETAILED DESCRIPTION:
The purpose of this study is to determine if local application of a commercially-available, FDA-approved preparation of enamel-matrix protein derivatives is effective in increasing clinical attachment levels (primary outcome), as well as alveolar bone (secondary outcome) compared to standard mechanical therapy in patients on periodontal maintenance therapy (PMT). Subjects will be divided into two groups for additional therapy in a 6-9 mm interproximal periodontal pocket at baseline: 1) local anesthesia and mini-flap reflection with subgingival mechanical debridement plus application of the enamel matrix protein derivate or 2) local anesthesia and mini-flap reflection with subgingival mechanical debridement plus application of saline. Samples/measurements will be obtained at the designated experimental site at baseline, 2 weeks, 6 and 12 months during PMT: 1) digital radiograph (baseline and 12 months only; bone height measurements), 2) presence of explorer-detectable supragingival plaque, 3) 30-second gingival crevicular fluid (GCF) sample (markers of inflammation, bone turnover), 4) recession from the cemento-enamel junction, 5) probing pocket depth and bleeding on probing (BOP). Following the 12-month visit, the research-specific interventions and measurements in the experimental quadrant will be removed from routine PMT.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic advanced adult periodontitis
* one quadrant with at least one 6-9 mm interproximal pocket
* overall good systemic health
* willingness to sign consent form

Exclusion Criteria:

* systemic diseases which significantly impact periodontal inflammation and bone turnover (e.g. rheumatoid arthritis)
* taking drugs which significantly impact periodontal inflammation and bone turnover
* surgical periodontal therapy within the past year
* pregnant or breast-feeding females

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Levels | 12 months
  This study is to determine if local application of a commercially-available, FDA-approved preparation of enamel-matrix protein derivatives is effective in increasing clinical attachment levels (periodontal tissue support) compared to standard mechanical therapy in patients on periodontal maintenance therapy (PMT). The following will be used in combination to evaluate impacts: digital radiograph (bone height), explorer-detectable supragingival plaque, 30-second GCF sample (markers of inflammation and bone turnover), recession, probing pocket depth (measurement of clinical attachment loss), and bleeding on probing (BoP).

SECONDARY OUTCOMES:
Alveolar bone | 12 months
  This study is to determine if local application of a commercially-available, FDA-approved preparation of enamel-matrix protein derivatives is effective in increasing alveolar bone compared to standard mechanical therapy in patients on periodontal maintenance therapy (PMT). The following will be used in combination to evaluate impacts: digital radiograph (bone height), explorer-detectable supragingival plaque, 30-second GCF sample (markers of inflammation and bone turnover), recession, probing pocket depth (measurement of clinical attachment loss), and bleeding on probing (BoP).

CONTACTS AND LOCATIONS:
Overall Officials: Amy Killeen, DDS, MS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, College of Dentistry, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No